CLINICAL TRIAL: NCT06548295
Title: Effects of Modified Constraint Induced Movement Therapy (mCIMT) Versus Conservative Treatment on Upper Extremity Motor Function and ADLs in Chronic Stroke Patients
Brief Title: Effects of mCIMT vs CT on Upper Extremity Motor Function and ADLs in Chronic Stroke Patients
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MSRSW/Batch-Fall22/733
Record Dates: First submitted 2024-08-07; First posted 2024-08-12 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Chronic Stroke
MeSH Terms: interventions — Conservative Treatment

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- modified constraint induced movement therapy (mCIMT) (Experimental)
  Interventions: Behavioral: modified constraint induced movement therapy (mCIMT)
- conservative treatment (Experimental)
  Interventions: Combination Product: conservative treatment

INTERVENTIONS:
Behavioral: modified constraint induced movement therapy (mCIMT) — Restraint the involved extremity by using a mitten. Repetitive task practice i.e filling a glass, drinking a glass of water, and eating with a spoon , stacking cones and stacking blocks, grasping and releasing of an object, reaching forward and sideways, lifting and dropping of an object from the one end of table to the other end.
  The shaping exercises included cube stacking, card turning, throwing balls into a box, grasping/holding and placing objects of different sizes, and drawing and painting exercises. Intervention: 5 sessions per week for 50 minutes for 6 weeks
  Arms: modified constraint induced movement therapy (mCIMT)
Combination Product: conservative treatment — The conservative rehabilitation program consisted of upper-limb range of motion exercises, positioning, stretching, and strengthening exercises, Passive mobilization of the shoulder ,elbow , wrist and small joints of hand Stretching of the affected arm including biceps, triceps and muscles of forearm and hand.
  Strengthening exercises of upper arm and forearm muscles involved. Intervention: 5 sessions per week for six weeks and 50 mintues
  Arms: conservative treatment

SUMMARY:
"Cerebral palsy (CP) affects gross motor function variably, with the spastic type notably impacting movement, coordination, and balance. Research highlights that spastic CP, characterized by muscle stiffness, can severely hinder activities like walking and running.

DETAILED DESCRIPTION:
Interventions such as gait training and vibrational therapy have shown promise in enhancing muscle function and body movements. A new device, EKKO, uses vibrational waves based on Neurotransmission Cognitive Theory to improve gross motor skills in children with CP by applying mechanical vibrations to nerve points. This study aims to compare the efficacy of EKKO therapy with traditional conservative treatments (such as range of motion exercises and balance training) in improving gross motor function in children with CP. Conducted over six months with randomized controlled trials, the research seeks to provide evidence-based insights into optimizing rehabilitation strategies for better motor performance and quality of life for CP patients.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be under the age of 40-75 years
* Diagnosis: stroke

Exclusion Criteria:

* patients suffering from motor dysfunction due to other diseases (e.g., cerebral palsy, traumatic brain injury, and Parkinson's disease
* Balance problem
* Rheumatic diseases
* High spasticity

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Barthal index | 12 Months
  Barthel Index (BI) stands out as a widely utilized measure for assessing basic activities of daily living (ADL). Scores of 0-20 indicate "total" dependency. Scores of 21-60 indicate "severe" dependency. Scores of 61-90 indicate "moderate" dependency.
The use of FMA-UE | 12 months
  measureing comprising 30 items for motor function and 3 items for reflex function, provides a comprehensive evaluation of motor abilities .
  In regards to UE feature, 33 elements evaluate motor function, six items assess sensitivity and proprioception, while the last 24 points rate joint pain and mobility.
  Every item of the assessment scale is marked on an ordinal level, from 0 to 2; the 0 value corresponds with the impossibility to perform a movement, and 2 represents the ability to perform a complete and adequate movement

CONTACTS AND LOCATIONS:
Locations (1):
- Little angles home aziz bhati shaheed road opposit junior aps, Sialkot, Pakistan

IPD SHARING:
Plan to Share IPD: No